CLINICAL TRIAL: NCT00481507
Title: Measuring the Influence of Kefir on Children's Stools on Antibiotics (MILK)
Acronym: MILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Lifeway Foods, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007-146
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Tract Infections
Keywords: Probiotic; Cultured dairy drink; Health; 10 day antibiotic; Otherwise healthy
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Kefir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Kefir (Experimental)
  Interventions: Other: Kefir

INTERVENTIONS:
Other: Kefir — The intervention was Kefir,a drink that is commercially available in the United States. The following probiotics are present in the Kefir: Lactococcus lactis, Lactococcus plantarum, Lactococcus rhamnosus, Lactococcus casei, Lactococcus lactis subspecies diacetylactis, Leuconostoc cremoris, Bifidobacterium longum, Bifidobacterium breve, Lactobacillus acidophilus, and 1 yeast, Saccharomyces florentinus. Parents were asked to ensure that their enrolled child consumed at least half of the bottle (150mL) everyday.
  Arms: Kefir
Other: Placebo — The intervention was Kefir, a drink that is commercially available in the United States. The following probiotics are present in active Kefir: Lactococcus lactis, Lactococcus plantarum, Lactococcus rhamnosus, Lactococcus casei, Lactococcus lactis subspecies diacetylactis, Leuconostoc cremoris, Bifidobacterium longum, Bifidobacterium breve, Lactobacillus acidophilus, and 1 yeast, Saccharomyces florentinus. The placebo group was heat-treated to kill all cultures. Parents were asked to ensure that their enrolled child consumed at least half of the bottle (150 mL)everyday.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of commercially available kefir on preventing antibiotic-associated diarrhea compared to placebo in children ages 1-5.

DETAILED DESCRIPTION:
Diarrhea is a common and costly disease of children in the United States. Children less than 5 years of age experience 20-35 million episodes of diarrhea per year. These episodes lead to 2-3.5 million physician visits (which account for 10% of all visits), more than 200,000 hospitalizations (13% of hospital admissions in children less than 5 years), and 325-425 deaths annually. In 1991, the outpatient costs of treating diarrhea for children under age 3 were calculated at 0.6-1 billion dollars per year.

Acute diarrhea in young children is almost always caused by infections or antibiotics. The rate of diarrhea associated with antibiotic usage is 20-35%, with children 3-36 months receiving on average 2-3 antibiotic prescriptions per year. Studies have shown that diarrhea due to either antibiotics or infections is caused by disturbances of the microflora of the gastrointestinal tract.

The current treatment for diarrhea in young children is oral rehydration, which is used to treat dehydration but plays no role in prevention. Probiotics are live microorganisms which, when administered in sufficient amounts, may improve health. Probiotics have the potential to treat and prevent diarrhea by improving the intestinal flora when disturbed by events such as antibiotics. Important to their use is that they are of human origin, survive passage through the gut, and are safe in very large dosages.

Studies have examined the potential health benefits of probiotics in the prevention and treatment of both antibiotic and infectious diarrhea. The probiotics have generally been given as supplements or pills. In placebo controlled randomized studies using these techniques, probiotics have generally been shown to decrease antibiotic associated diarrhea by 15-25% over placebo. Other studies have enrolled children with acute diarrhea, generally from rotavirus, and found a 30-50% cure rate in the probiotic group over placebo.

Kefir, available in the United States, is a milk product derived by the action of ten probiotics. A daily dose of 10^6-10^9 colony forming units of probiotics has been studied and recommended for health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and write English
* Aged 1-5 years
* Male or female
* Diagnosed with an upper respiratory infection and placed on a penicillin class antibiotic regimen for 10 days

Exclusion Criteria:

* Developmental delays
* Chronic conditions, such as diabetes or asthma, that require medication
* Prematurity, birth weight <2500 grams
* Allergy to kefir and/or milk
* Active diarrhea
* Congenital anomalies
* Failure to thrive
* Parental belief of lactose intolerance

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2007-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Merenstein, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Deptartment of Family Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Merenstein DJ, Foster J, D'Amico F. A randomized clinical trial measuring the influence of kefir on antibiotic-associated diarrhea: the measuring the influence of Kefir (MILK) Study. Arch Pediatr Adolesc Med. 2009 Aug;163(8):750-4. doi: 10.1001/archpediatrics.2009.119. PMID 19652108

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 150mL per day, administered orally for 10 consecutive days. Placebo was heat-treated to kill all cultures.
- Kefir: 150mL per day, administered orally for 10 consecutive days. Active kefir contained probiotics Lactococcus lactis, Lactococcus plantarum, Lactococcus rhamnosus, Lactococcus casei, Lactococcus lactis subspecies diacetylactis, Leuconostoc cremoris, Bifidobacterium longum, Bifidobacterium breve, Lactobacillus acidophilus, and 1 yeast, Saccharomyces florentinus.
Period: Overall Study
Arm/Group | Placebo | Kefir
Started | 64 | 61
Completed | 64 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Kefir | Total
Number analyzed (Participants) | 64 | 61 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 61 | 125
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 31 | 33 | 64
Region of Enrollment [Number; unit: participants]
  United States | 64 | 61 | 125

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Participants With Diarrhea by Parental Report
Description: The primary outcome was the incidence of participants receiving antibiotics with diarrhea during the 14-day follow-up period, as determined by parental report.
Time Frame: 14 days
Population: Prior estimates of the sample size showed that 62 per group would have 80% power for detecting a difference of 20% in the rates of diarrhea. This was based on the placebo group having a 10% (which is consistent with published literature) rate of diarrhea. Analysis performed used the intention to treat and no imputation was required.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Kefir | Placebo
Number analyzed (Participants) | 61 | 64
Percentage of participants | 18.0 [9 to 30] | 21.9 [13 to 24]
Statistical Analysis 1: Comparison: Kefir vs Placebo; Reply: The null hypothesis was the rates of diarrhea for Kefir vs. Placebo are not different. Post power calculation was not performed because the difference observed (21.9% vs. 18%) was less than a difference that which would be considered clinically important; Test type: Superiority or Other; p > .05, Chi-squared — Reply: Only one test was performed for the primary outcome. No covariates were entered into this model and p-value is unadjusted; The results obtained from the logistic regression are equivalent to the chi-square test with one degree of freedom; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.54 to 1.43]

2. Secondary Outcome: Incidence of Vomiting, Stomach Pain, Constipation, Runny Nose, Cough, Earaches, Fever, Irritability, Lethargy, and Loose Stools
Description: Incidence of Vomiting, Stomach Pain, Constipation, Runny Nose, Cough, Earaches, Fever, Irritability, Lethargy, and Loose Stools. Outcomes assessed by parental report via daily diary and phone follow-ups with study research assistants on days 0, 5, 10, and 15.
Time Frame: 14 days
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Kefir | Placebo
Number analyzed (Participants) | 61 | 64
Percentage of participants
  vomiting | 16.4 [8 to 28] | 10.9 [5 to 21]
  stomach pain | 8.2 [3 to 18] | 14.1 [7 to 25]
  constipation | 19.7 [11 to 32] | 17.2 [9 to 29]
  runny nose | 77.0 [65 to 87] | 82.8 [71 to 91]
  cough | 68.9 [56 to 80] | 53.1 [40 to 66]
  earaches | 23.0 [13 to 36] | 17.2 [9 to 29]
  fever | 45.9 [33 to 59] | 39.1 [27 to 52]
  irritability | 19.7 [11 to 32] | 18.8 [10 to 31]
  lethargy | 16.4 [8 to 28] | 21.9 [13 to 46]
  loose stools | 29.5 [19 to 43] | 32.8 [22 to 46]

ADVERSE EVENTS:
Arm/Group | Placebo | Kefir
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/61
Other Adverse Events (participants affected / at risk) | 1/64 | 1/61
OTHER ADVERSE EVENTS (reported when occurring in more than 1.6% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Kefir (N=61)
emesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
We did not assess or culture stools for the presence of pathogenic organisms. We did not independently examine children; we relied on parental/patient-oriented outcomes. Our population was generally very healthy. We did not assess probiotic dosages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No